CLINICAL TRIAL: NCT03888430
Title: Transcutaneous PCO2 Assessment During Intubation in ICU
Acronym: C-TOP
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3030_C-TOP
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Intubation in ICU
Keywords: Transcutaneous PCO2; Preoxygenation; Post-intubation hypotension; ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard Oxygen: preoxygenation methods : Standard Oxygen
  Interventions: Procedure: PtcCO2 measure during intubation
- High flow Oxygen: preoxygenation methods : High flow Oxygen
  Interventions: Procedure: PtcCO2 measure during intubation
- Non invasive ventilation: preoxygenation methods : Non invasive ventilation
  Interventions: Procedure: PtcCO2 measure during intubation

INTERVENTIONS:
Procedure: PtcCO2 measure during intubation — Transcutaneous measure during intubation. Non invasive measure without any risk according to the literature

SUMMARY:
PtcCO2 assessement during intubation in ICU. Comparison of three different preoxygenation methods.

DETAILED DESCRIPTION:
Transcutaneous PCO2 assessement during intubation in ICU. Comparison of three different preoxygenation methods and hemodynamic changes during this period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years of age or older
* Requiring intubation in Resuscitation

Exclusion Criteria:

* Contraindication to orotracheal intubation
* Intubation in a respiratory or cardiocirculatory arrest situation
* Need for intubation in great urgency preventing the installation of the transcutaneous capnia sensor and its calibration
* Major Incapable
* Opposition of the patient or his relatives to the research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU patients requiring intubation
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-04-13 (Actual)

PRIMARY OUTCOMES:
Transcutaneous carbon dioxide partial pressure variation during intubation | 4 hours after intubation (the day of inclusion)
  Transcutaneous carbon dioxide partial pressure (TcPO2) variation during intubation in ICU and within 4 hours after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien FREROU, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France